CLINICAL TRIAL: NCT00114777
Title: Belatacept Evaluation of Nephroprotection and Efficacy as First-line Immunosuppression Trial - Extended Criteria Donors (BENEFIT-EXT)
Brief Title: Study of Belatacept in Subjects Who Are Undergoing a Renal Transplant
Acronym: BENEFIT-EXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IM103-027
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cyclosporin A (Active Comparator)
  Interventions: Drug: Cyclosporin A
- Belatacept Less Intensive Regimen (LI) (Experimental)
  Interventions: Drug: Belatacept Less Intensive Regimen (LI)
- Belatacept More Intensive Regimen (MI) (Experimental)
  Interventions: Drug: Belatacept More Intensive Regimen (MI)

INTERVENTIONS:
Drug: Cyclosporin A — tablet, oral, 1st month target: 150-300 ng/mL, after 1st month target: 100-250 ng/mL, daily, 36 months, 100-250 ng/mL, daily, 84 months
  Other Names: CsA
  Arms: Cyclosporin A
Drug: Belatacept Less Intensive Regimen (LI) — solution, IV, 10mg/kg: Days 1 and 5, Weeks 2, 4, 8 and 12, then 5 mg/kg every 4 weeks, q 4 weeks, 36 months months, 5 mg/kg every 4 weeks, q 4 weeks, 84 months
  Arms: Belatacept Less Intensive Regimen (LI)
Drug: Belatacept More Intensive Regimen (MI) — solution, IV, 10mg/kg: Days 1 and 5, Weeks 2, 4, 6, 8, 10,12, 16, 20, and 24, then 5 mg/kg every 4 weeks, q 4 weeks, 36 months, 5 mg/kg every 4 weeks, q 4 weeks, 84 months
  Arms: Belatacept More Intensive Regimen (MI)

SUMMARY:
The purpose of this trial is to learn if Belatacept is effective and safe as a first line of immunosuppression treatment in patients undergoing a renal transplant where the donor kidney is obtained in patients with extended criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a first-time recipient of a kidney transplant from a deceased donor.
* Specific donor criteria

Exclusion Criteria:

* Donor age <10 years
* Subjects receiving a concurrent solid organ or cell transplant (lung, heart, etc.)
* Subjects with a positive T-cell lymphocytotoxic crossmatch.
* Subjects who are positive for Hepatitis B or C, or HIV
* Active tuberculosis
* History of cancer in the last 5 years
* History of substance abuse
* Specific laboratory results are exclusionary
* Mammography suspicious for cancer
* Allergy to iodine
* For Long-term extension study-Subjects who have completed three years of study treatment (through Week 156)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2005-02; Primary Completion 2008-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (74):
- United States (28):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Ucla Kidney & Kidney-Pancreas Transplant Research Office, Los Angeles, California
  - National Institute Of Transplantation, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - University Of California San Francisco Medical Center, San Francisco, California
  - University Of Colorado Health Sciences Center, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Lifelink Healthcare Institute, Tampa, Florida
  - Piedmont Transplant Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University-Feinberg School Of Medicine, Chicago, Illinois
  - University Of Chicago Hospitals, Chicago, Illinois
  - Acadiana Renal Physicians, New Iberia, Louisiana
  - Tulane Abdominal Transplant Institute, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Western New England Renal & Transplant Associates, Pc, Springfield, Massachusetts
  - Henry Ford Hospital, Transplant Institute, Detroit, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Mount Sinai School Of Medicine, New York, New York
  - Columbia University College Of Physicians & Surgeons, New York, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Drexel University College Of Medicine, Department Of Surgery, Philadelphia, Pennsylvania
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University Of Wisconsin, Madison, Wisconsin
  - Froedtert Memorial Hospital, Milwaukee, Wisconsin
- Argentina (4):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Cordoba, Crd, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Santa Fe
- Local Institution, Woodville, South Australia, Australia
- Austria (2):
  - Local Institution, Innsbuck
  - Local Institution, Vienna
- Local Institution, Leuven, Belgium
- Brazil (5):
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre/rs, Rio Grande do Sul
  - Local Institution, Campinas/sp, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Montreal, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Local Institution, Prague, Czechia
- France (9):
  - Local Institution, Bordeaux
  - Local Institution, Brest
  - Local Institution, Créteil
  - Local Institution, Le Kremlin-Bicêtre
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Toulouse
  - Local Institution, Tours
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Hanover
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Szeged
- Italy (3):
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Roma
- Local Institution, Oslo, Norway
- Poland (2):
  - Local Institution, Poznan
  - Local Institution, Warsaw
- Local Institution, Pretoria, Gauteng, South Africa
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Málaga
- Local Institution, Gothenburg, Sweden
- Local Institution, Manchester, United Kingdom

REFERENCES:
- [Derived] Dobbels F, Wong S, Min Y, Sam J, Kalsekar A. Beneficial effect of belatacept on health-related quality of life and perceived side effects: results from the BENEFIT and BENEFIT-EXT trials. Transplantation. 2014 Nov 15;98(9):960-8. doi: 10.1097/TP.0000000000000159. PMID 24831918
- [Derived] Pestana JO, Grinyo JM, Vanrenterghem Y, Becker T, Campistol JM, Florman S, Garcia VD, Kamar N, Lang P, Manfro RC, Massari P, Rial MD, Schnitzler MA, Vitko S, Duan T, Block A, Harler MB, Durrbach A. Three-year outcomes from BENEFIT-EXT: a phase III study of belatacept versus cyclosporine in recipients of extended criteria donor kidneys. Am J Transplant. 2012 Mar;12(3):630-9. doi: 10.1111/j.1600-6143.2011.03914.x. Epub 2012 Feb 2. PMID 22300431
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 595 participants enrolled, 578 randomized. Reasons for non-randomization included 13 subjects no longer met study criteria; 3 discontinued on sponsor's discretion; 1 due to other reason. Of those randomized, 543 were treated. Reasons for non-treatment were not specified.
Groups:
- Belatacept More Intensive (MI) Regimen: Belatacept 10 mg/kg intravenous solution on Days 1 and 5 during the first week, and then every other week through 3 months (Weeks 2, 4, 8, and 12) and then every 4 weeks through 6 months (Weeks 16, 20 and 24), followed by a maintenance dose of belatacept, 5 mg/kg intravenously every 4 weeks thereafter for up to 84 months
- Belatacept Less Intensive (LI) Regimen: Belatacept 10 mg/kg intravenously on Day 1 and Day 5 during the first week, and then every other week for 4 weeks (Weeks 2 and 4), and then every 4 weeks for 2 months (Weeks 8 and 12), followed by a maintenance dose of belatacept, 5 mg/kg intravenously every 4 weeks thereafter for up to 84 months.
- Cyclosporin A (CsA): Cyclosporin A 4-10 mg/kg capsules orally in 2 divided doses, adjusted thereafter to maintain serum concentrations of 150-300 ng/mL during the first month. Subsequently, doses were adjusted to maintain a predefined range of trough serum concentrations of 100-250 ng/mL for up to 84 months.
Period: Randomization to Month 36
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Started | 184 | 175 | 184
Completed | 109 | 114 | 100
Not Completed | 75 | 61 | 84
Not completed — Death | 10 | 4 | 3
Not completed — No Longer Met Study Criteria | 0 | 0 | 2
Not completed — Lack of Efficacy | 19 | 15 | 17
Not completed — Poor or Non-Compliance | 0 | 0 | 1
Not completed — Adverse Event | 34 | 35 | 44
Not completed — Withdrawal by Subject | 3 | 4 | 5
Not completed — Other | 9 | 3 | 12
Period: Long-Term Extension to Month 84
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Started | 104 | 113 | 87
Completed | 74 | 84 | 57
Not Completed | 30 | 29 | 30
Not completed — Death | 8 | 13 | 7
Not completed — No Longer Met Study Criteria | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Poor or Non-Compliance | 1 | 1 | 3
Not completed — Adverse Event | 15 | 14 | 7
Not completed — Withdrawal by Subject | 2 | 1 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Administrative Reason by Sponsor | 0 | 0 | 1
Not completed — Other | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Belatacept More Intensive (MI) Regimen: Belatacept 10mg/kg intravenous solution for over 30 minutes on Day 1 and 5 of Week 2, 4, 6, 8, 10, 12, 16, 20, and 24 and 5mg/kg intravenous solution for over 30 minutes every 4 weeks up to 84 months.
- Belatacept Less Intensive (LI) Regimen: Belatacept 10mg/kg intravenous solution for over 30 minutes on Day 1 and 5 of Week 2, 4, 8, 12 followed by belatacept 5mg/kg intravenous solution every 4 weeks up to 84 months.
- Cyclosporin A (CsA): Cyclosporine A 410 mg/kg was capsules, orally, twice daily in 2 divided dose for 1 month, to maintain serum concentration of 150-300 ng/mL. The subsequent dose was adjusted to maintain a predefined range of trough serum concentrations of 100-250/mL, daily for up to 84 months.
- Total: Total of all reporting groups
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA) | Total
Number analyzed (Participants) | 184 | 175 | 184 | 543
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (12.6) | 56.1 (12.4) | 55.7 (12.2) | 56.2 (12.4)
Age, Customized [Number; unit: participants]
  18 to 45 years | 32 | 35 | 34 | 101
  46 to 65 years | 100 | 97 | 108 | 305
  more than 65 years | 52 | 43 | 42 | 137
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 46 | 68 | 179
  Male | 119 | 129 | 116 | 364

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Survived With a Graft at 12 Months Post-Transplant
Description: Participant and graft survival at 12 months was summarized within each treatment group. Graft loss was defined as either functional loss or physical loss (nephrectomy). Functional loss was defined as a sustained level of serum creatinine ≥ 6.0 mg/dL (530 μmol/L) as determined by central laboratory for ≥4 weeks or 56 or more consecutive days of dialysis.
Time Frame: Month 12 post-transplant
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cyclosporin A (CsA): Cyclosporin A 410 mg/kg capsules, orally, twice daily in 2 divided dose for 1 month, to maintain serum concentration of 150-300 ng/mL. The subsequent dose was adjusted to maintain a predefined range of trough serum concentrations of 100-250/mL, daily for up to 84 months.
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants | 85.9 [80.8 to 90.9] | 88.0 [83.2 to 92.8] | 84.8 [79.6 to 90.0]
Statistical Analysis 1: Comparison: Belatacept More Intensive (MI) Regimen vs Cyclosporin A (CsA); Test type: Superiority or Other; Treament Difference = 1.1, 97.3% CI 2-sided [-7.2 to 9.4] — The treatment differences between each belatacept treatment group and cyclosporin group was tested at the 0.027 significance level for participant and graft survival (based on 10% non-inferiority margin)
Statistical Analysis 2: Comparison: Belatacept Less Intensive (LI) Regimen vs Cyclosporin A (CsA); Test type: Superiority or Other; Treatment difference = 3.2, 97.3% CI 2-sided [-5.0 to 11.4] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants With a Measured Glomerular Filtration Rate (GFR) <60 mL/Min Per 1.73 m^2 at Month 12 or a Decrease in Measured GFR >=10 mL/Min Per 1.73 m^2 From Month 3 to Month 12
Description: GFR was assessed using a true measure of glomerular filtration via non-radiolabeled iothalamate clearance test using a validated procedure.
Time Frame: From Month 3 to Month 12
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants
  Measured GFR <60 mL/min/1.73 m^2 (Month 12) | 55.7 [48.3 to 63.0] | 62.1 [54.8 to 69.4] | 67.4 [60.5 to 74.3]
  GFR ≥ 10 mL/min/1.73 m^2 (Month 3 to Month 12) | 17.6 [12.0 to 23.2] | 27.2 [20.5 to 33.9] | 24.7 [18.4 to 31.1]
Statistical Analysis 1: Comparison: Belatacept More Intensive (MI) Regimen vs Cyclosporin A (CsA); Test type: Superiority or Other; p = 0.0018, Chi-squared; Percentage difference = -14.4, 97.3% CI 2-sided [-24 to -4.7] — A continuity-corrected chi-squared test at the significance level 0.027 was performed to assess the effect of each belatacept regimen compared with cyclosporin A
Statistical Analysis 2: Comparison: Belatacept Less Intensive (LI) Regimen vs Cyclosporin A (CsA); Test type: Superiority or Other; p = 0.0616, Chi-squared; Percentage difference = -8.5, 97.3% CI 2-sided [-18 to 0.9] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Measured Glomerular Filtration Rate (GFR) by Month 12 and 24
Description: GFR was assessed using a true measure of glomerular filtration via nonradiolabeled iothalamate clearance test using a validated procedure. Missing measured GFR assessments were imputed. Here, 'n' signifies the number of evaluable participants for the reporting arm at the given time point. Missing measured GFR assessments were imputed to a GFR of zero.
Time Frame: At Month 12 and Month 24
Population: All randomized and transplanted participants
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
mL/min/1.73 m^2
  Month 12 (n = 154,151,154) | 52.1 (21.9) | 49.5 (25.4) | 45.2 (21.1)
  Month 24 (n = 136,139,136) | 51.5 (22.9) | 49.7 (23.67) | 45.0 (27.18)

4. Secondary Outcome: Percentage of Participants With Chronic Allograft Nephropathy (CAN) at Month 12
Description: Biopsy-proven CAN was determined by a blinded central histopathologist using the Banff 97 working classification of kidney transplant pathology. Onset of CAN was determined by the biopsy date when it was observed. Participants were considered as having CAN at 12 months if: CAN observed in a biopsy either prior to 12 months (including baseline biopsy) or first post 12 months biopsy; Participant had graft loss during the first year post transplant; no biopsy available post 12 months and CAN not observed in biopsies prior to 12 months; no biopsy available either prior to or post 12 months; and the measured glomerular filtration rate from Month 3 to Month 12 decreases at least 10 mL/min/1.73m^2. All other participants with missing 12 month biopsy were considered having no CAN observed at 12 months.
Time Frame: At Month 12
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants | 44.8 [37.6 to 52.0] | 46.0 [38.6 to 53.4] | 51.6 [44.4 to 58.9]

5. Secondary Outcome: Percentage of Participants Who Survived With a Graft at 24 and 36 Months Post-Transplant
Description: Participant and graft survival at 12 months was summarized within each treatment group. Graft loss was defined as either functional loss or physical loss (nephrectomy). Functional loss will be defined as a sustained level of serum creatinine ≥ 6.0 mg/dL (530 μmol/L) as determined by central laboratory for ≥ 4 weeks or 56 or more consecutive days of dialysis.
Time Frame: Month 24 and Month 36 post-transplant
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants
  Month 24 | 82.6 [77.1 to 88.1] | 84.0 [78.6 to 89.4] | 82.6 [77.1 to 88.1]
  Month 36 | 80.4 [74.7 to 86.2] | 82.3 [76.6 to 87.9] | 79.9 [74.1 to 85.7]

6. Secondary Outcome: Calculated Glomerular Filtration Rate (GFR) at 6, 12, 24, 36 and 84 Months
Description: GFR was assessed using a true measure of glomerular filtration via nonradiolabeled iothalamate clearance test using a validated procedure. Missing measured GFR assessments were imputed. Here 'n' signifies those participants evaluable for this measure at specified time points for each arm, respectively.
Time Frame: Months 6, 12, 24, 36 and 84
Population: All randomized and transplanted participants
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
participants
  Month 6 (n = 161,152,153) | 43.6 (21.67) | 43.4 (18.57) | 35.5 (20.51)
  Month 12 (n = 159,154,154) | 44.4 (22.78) | 44.8 (21.57) | 36.5 (21.08)
  Month 24 (n = 152,158,154) | 44.4 (26.72) | 42.8 (24.07) | 34.9 (21.59)
  Month 36 (n = 152,154,143) | 42.7 (27.59) | 42.2 (25.2) | 31.5 (22.13)
  Month 84 (n = 69,79,51) | 57.6 (18.58) | 59.1 (18.85) | 44.6 (17.37)

7. Secondary Outcome: Change in Calculated GFR at Months 12, 24, 36 and 84
Description: as for outcome 6
Time Frame: Baseline and Months 12, 24, 36 and 84
Population: All randomized and transplanted participants
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
mL/min/1.73 m^2
  Month 12 (n = 159,154,154) | -0.7 (17.96) | -0.6 (15.39) | -1.1 (12.48)
  Month 24 (n = 146,154,149) | -1.4 (17.68) | -1.6 (18.7) | -3.6 (15.37)
  Month 36 (n = 146,150,139) | -2.9 (23.7) | -2.1 (20.92) | -6.1 (17.39)
  Month 84 (n = 67,76,49) | 7.5 (17.48) | 10.4 (17.54) | -4.0 (17.17)

8. Secondary Outcome: Number of Participants With Anti-Hypertensive Medications Used to Control Hypertension at 12, 24 and 36 Months
Description: Participants were determined to have hypertension at a particular time point if standardized systolic blood pressure ≥ 130 mm Hg or standardized diastolic blood pressure ≥ 80 mm Hg or participant had received an antihypertensive medication(s) for hypertension. Here 'n' signifies those participants evaluable for this measure at specified time points for each arm, respectively.
Time Frame: Baseline and Months 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
participants
  1-2 Medications at Month 12 (n=184,175,184) | 82 | 79 | 76
  ≥ 3 Medications at Month 12 (n=184,175,184) | 76 | 66 | 93
  1-2 Medications at Month 24 (n=177,170,179) | 80 | 79 | 71
  ≥ 3 Medications at Month 24 (n=177,170,179) | 78 | 65 | 89
  1-2 Medications at Month 36 (n=151,145,143) | 65 | 67 | 51
  ≥ 3 Medications at Month 36 (n=151,145,143) | 70 | 60 | 79

9. Secondary Outcome: Percentage of Subjects Who Used Anti-Hypertensive Medications to Control Hypertension at Months 12, 24 and 36
Description: Participants were determined to have hypertension at a particular time point if standardized systolic blood pressure ≥ 130 mm Hg or standardized diastolic blood pressure ≥ 80 mm Hg or subject had received an anti-hypertensive medication(s) for hypertension. Here 'n' signifies those participants evaluable for this measure at specified time points for each arm, respectively.
Time Frame: Months 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants
  Month 12 (n = 184,175,184) | 87 [82.09 to 91.82] | 83.4 [77.92 to 88.94] | 87.0 [82.09 to 91.82]
  Month 24 (n = 177,170,179) | 89.3 [84.71 to 93.83] | 84.7 [9.3 to 90.12] | 89.4 [84.87 to 93.9]
  Month 36 (n = 151,145,143) | 89.4 [84.49 to 94.31] | 87.6 [82.22 to 92.25] | 90.9 [86.2 to 95.62]

10. Secondary Outcome: Percentage of Participants With New Onset Diabetes Mellitus (NODM) at 12, 24 and 36 Months.
Description: NODM was defined as participant who did not have diabetes prior to randomization. Participants were determined for NODM if the participant received an antidiabetic medication for a duration of at least 30 days, or at least two fasting plasma glucose (FPG) tests indicate that FPG is ≥ 126 mg/dL (7.0 mmol/L).
Time Frame: Months 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants
  12 Month | 2.3 [0.2 to 5.4] | 5.1 [1.4 to 8.9] | 9.3 [4.1 to 14.6]
  24 Month | 3.0 [0.8 to 7.6] | 7.4 [3.0 to 11.7] | 9.3 [4.1 to 14.6]
  36 Month | 5.3 [1.5 to 9.1] | 9.6 [4.6 to 14.5] | 9.3 [4.1 to 14.6]

11. Secondary Outcome: Systolic and Diastolic Blood Pressure (BP) at 12, 24 and 36 Months
Description: Participants were determined to have hypertension at a particular time point if standardized systolic blood pressure ≥ 130 mm Hg or standardized diastolic blood pressure ≥ 80 mm Hg or participant had received an anti-hypertensive medication(s) for hypertension. Here 'n' signifies those participants evaluable for this measure at specified time points for each arm, respectively.
Time Frame: Months 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
mmHg
  Diastolic BP (Month 12) (n= 184,175,184) | 77.8 (13.83) | 78.3 (10.62) | 81.8 (11.68)
  Systolic BP (Month 12) (n= 184,175,184) | 141.4 (21.29) | 140.9 (21.09) | 149.5 (19.81)
  Diastolic BP (Month 24) (n= 120,129,120) | 78.2 (13.28) | 77.0 (11.18) | 81.7 (11.47)
  Systolic BP (Month 24) (n= 120,129,120) | 138.82 (24.31) | 136.7 (20.96) | 146.8 (21.11)
  Diastolic BP (Month 36) (n= 112,119,108) | 75.4 (11.55) | 75.2 (10.85) | 77.2 (11.79)
  Systolic BP (Month 36) (n= 112,119,108) | 134.9 (19.54) | 134.7 (21.59) | 140.7 (21.19)

12. Secondary Outcome: Mean Framingham Risk Score From Baseline to Months 12, 24 and 36
Description: The risk score was calculated based on the total points from six variables: Age, Level of LDL-cholesterol, Level of HDL-cholesterol, Presence and severity of systolic or diastolic hypertension, Presence or absence of a history of diabetes mellitus and Presence or absence of a history recent cigarette smoking. Total scores can range from <-3 to >14, which translate to a 1% to 56% risk of developing coronary heart disease in 10 years. Totals in the 4 to 6 point range translate to a 7 to 11% risk and 8 to 10 point range translate to a 18 to 27% risk.
Time Frame: Baseline and Months 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Belatacept Less Intensive (LI) Regimen: Belatacept 10mg/kg intravenous solution for over 30 minutes on Day 1 and 5 of Week 2, 4, 8, 12 followed by belatacept 5mg/kg intravenous solution every 4 weeks up to 84months.
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
units on a scale
  Month 12 | 5.3 (4.11) | 4.5 (4.02) | 6.0 (3.98)
  Month 24 | 5.0 (4.25) | 4.6 (4.23) | 6.2 (4.07)
  Month 36 | 5.2 (4.18) | 4.9 (3.84) | 5.8 (4.00)

13. Secondary Outcome: Percentage of Participants Using Lipid-Lowering Therapy at 12, 24, and 36 Months
Description: Dyslipidemia was defined as triglyceride ≥ 500 mg/dL [5.65 mmol/L], low density lipoprotein (LDL) ≥ 100 mg/dL [2.59 mmol/L], and non-elevated high density lipoprotein (HDL) ≥ 130 mg/dL [3.36 mmol/L]. Here 'n' signifies those participants evaluable for this measure at specified time points for each arm, respectively.
Time Frame: Months 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants
  Month 12 (n=184.175,184) | 43.5 [36.3 to 50.6] | 40.0 [32.7 to 47.3] | 46.2 [39.0 to 53.2]
  Month 24 (n=184,175,184) | 47.8 [40.6 to 55.0] | 42.3 [35.0 to 49.6] | 51.1 [43.9 to 58.3]
  Month 36 (n=151,145,143) | 52.3 [44.4 to 60.3] | 45.5 [37.4 to 53.6] | 60.8 [52.8 to 68.8]

14. Secondary Outcome: Change in Total Cholesterol (TC), Non-HDL, LDL and HDL Cholesterol and Triglycerides at 12, 24 and 36
Description: Dyslipidemia was defined as triglyceride ≥ 500 mg/dL [5.65 mmol/L], low density lipoprotein (LDL) ≥ 100 mg/dL [2.59 mmol/L], and elevated non-high density lipoprotein (HDL) ≥ 130 mg/dL [3.36 mmol/L]. Here 'n' signifies those participants evaluable for this measure at specified time points for each arm, respectively.
Time Frame: Months 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
mg/dL
  Non-HDL (Month 12) (n=184,175,184) | 134.5 (45.04) | 134.2 (40.69) | 153.4 (46.99)
  TC (Month 12) (n =184,175,184) | 183.7 (47.72) | 184.1 (45.51) | 201.3 (49.49)
  Triglyceride (Month 12) (n=184,175,184) | 171.9 (129.76) | 153.2 (69.92) | 213.8 (113.12)
  HDL (Month 12) (n=184,175,184) | 49.2 (13.73) | 49.8 (15.85) | 47.9 (14.76)
  LDL (Month 12) (n=184,175,184) | 104.0 (39.33) | 102.4 (36.63) | 107.8 (40.08)
  Non--HDL (Month 24) (n=119,128,111) | 126.1 (45.45) | 129.8 (37.89) | 148.7 (60.46)
  TC (Month 24) (n=119,128,111) | 175.6 (47.99) | 178.0 (41.9) | 195.7 (61.46)
  Triglyceride (Month 24) (n=98,104,93) | 152.0 (108.97) | 147.0 (69.45) | 208.2 (135.19)
  HDL (Month 24) (n=119,128,111) | 49.5 (16.27) | 48.2 (14.41) | 47.0 (17.77)
  LDL (Month 24) (n=97,104,93) | 96.9 (33.46) | 101.4 (36.64) | 108.6 (40.8)
  Non-HDL (Month 36) (n=111,117,97) | 132.6 (41.86) | 132.2 (46.81) | 139.1 (49.68)
  TC (Month 36) (n=111,117,98) | 181.0 (43.84) | 181.9 (49.16) | 196.7 (127.35)
  Triglyceride (Month 36) (n=80,88,78) | 160.7 (98.56) | 154.3 (76.58) | 181.3 (108.32)
  HDL (Month 36) (n=111,117,97) | 48.9 (14.82) | 49.6 (16.24) | 47.0 (14.28)
  LDL (Month 36) (n=79,88,77) | 103.1 (32.59) | 106.0 (37.29) | 102.3 (47.4)

15. Secondary Outcome: Percentage of Participants Who Have an Acute Rejection by Months 6, 12, 24, 36 and 84
Description: Acute rejection was defined as central biopsy proven rejection that was either clinically suspected by protocol defined reasons or clinically suspected by other reasons and treated. Clinically suspected acute rejection was defined as an unexplained rise of serum creatinine ≥ 25% from baseline creatinine or an unexplained decreased urine output or fever and graft tenderness or serum creatinine that remains elevated within 14 days post--transplantation and clinical suspicion of acute rejection exists.
Time Frame: Months 6, 12, 24, 36 and 84
Population: All randomized and transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants
  Month 6 | 17.4 [11.9 to 22.9] | 16.6 [11.1 to 22.1] | 13.6 [8.6 to 18.5]
  Month 12 | 17.4 [11.9 to 22.9] | 17.7 [12.1 to 23.4] | 14.1 [9.1 to 19.2]
  Month 24 | 17.4 [11.9 to 22.9] | 18.3 [12.6 to 24.0] | 15.2 [10.0 to 20.4]
  Month 36 | 17.9 [12.4 to 23.5] | 18.9 [13.1 to 24.7] | 15.8 [10.5 to 21.0]
  Month 84 | 19.0 [13.4 to 24.7] | 19.4 [13.6 to 25.3] | 15.8 [10.5 to 21.1]

16. Secondary Outcome: Number of Participants Using Lymphocyte Depleting Therapy and Steroid-Resistant for Acute Rejection by Months 6, 12, 24, and 36.
Description: Acute rejection was defined as central biopsy proven rejection that was either clinically suspected by protocol defined reasons or clinically suspected by other reasons and treated. Lymphocyte -depletion therapy for treatment of an episode of acute was defined as a participant treated with therapy and provided not treated with steroids earlier while steroid resistant acute rejection was defined as participants initially treated with steroids alone for suspected acute rejection for at least 2 days and then followed by the start of lymphocyte -depletion therapy.
Time Frame: Months 6, 12, 24 and 36
Population: All randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
participants
  Only corticosteroid treated (Month 6) | 14 | 16 | 9
  Corticosteroid resistant (Month 6) | 2 | 2 | 2
  Lymphocyte-depleting treated (Month 6) | 13 | 5 | 4
  Only corticosteroid treated (Month 12) | 14 | 16 | 10
  Corticosteroid resistant (Month 12) | 2 | 2 | 2
  Lymphocyte-depleting treated (Month 12) | 13 | 5 | 4
  Only corticosteroid treated (Month 24) | 13 | 19 | 11
  Corticosteroid resistant (Month 24) | 2 | 1 | 2
  Lymphocyte-depleting treated (Month 24) | 14 | 7 | 4
  Only corticosteroid treated (Month 36) | 13 | 19 | 11
  Corticosteroid resistant (Month 36) | 2 | 1 | 2
  Lymphocyte-depleting treated (Month 36) | 14 | 7 | 4

17. Secondary Outcome: Number of Participants Based on Severity of Acute Rejection Based on Banff Grade Level by Months 6, 12, 24, 36 and 84
Description: as for outcome 15
Time Frame: Months 6, 12, 24, 36 and 84
Population: All randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
participants
  Mild acute (IA) (Month 6) | 0 | 4 | 2
  Mild acute (IB) (Month 6) | 6 | 2 | 2
  Moderate acute (IIA) (Month 6) | 11 | 15 | 16
  Moderate acute (IB) (Month 6) | 15 | 8 | 5
  Severe acute (III) (Month 6) | 0 | 0 | 0
  Mild acute (IA) (Month 12) | 0 | 4 | 2
  Mild acute (IB) (Month 12) | 6 | 2 | 2
  Moderate acute (IIA) (Month 12) | 11 | 17 | 17
  Moderate acute (IB) (Month 12) | 15 | 8 | 5
  Severe acute (III) (Month 12) | 0 | 0 | 0
  Mild acute (IA) (Month 24) | 0 | 4 | 2
  Mild acute (IB) (Month 24) | 6 | 2 | 3
  Moderate acute (IIA) (Month 24) | 10 | 17 | 18
  Moderate acute (IB) (Month 24) | 16 | 9 | 5
  Severe acute (III) (Month 24) | 0 | 0 | 0
  Mild acute (IA) (Month 36) | 0 | 4 | 2
  Mild acute (IB) (Month 36) | 6 | 2 | 4
  Moderate acute (IIA) (Month 36) | 10 | 18 | 18
  Moderate acute (IIB) (Month 36) | 16 | 9 | 5
  Severe acute (III) (Month 36) | 1 | 0 | 0
  Mild acute (IA) (Month 84) | 0 | 4 | 2
  Mild acute (IB) (Month 84) | 6 | 6 | 4
  Moderate acute (IIA) (Month 84) | 12 | 18 | 18
  Moderate acute (IIB) (Month 84) | 16 | 9 | 5
  Severe acute (III) (Month 84) | 1 | 0 | 0

18. Secondary Outcome: Mean Changes in Mental Component and Physical Component Health-Related Quality of Life (SF-36) From Baseline to Months 12, 24 and 36
Description: The SF-36 is a 36-item self-administered questionnaire developed to assess health-related quality of life (QOL) and comprises 8 domains, including 4 physical (physical health, bodily pain, physical functioning and physical role limitations) and 4 mental (mental health, vitality, social functioning, and emotional role limitation) subscales. Responses are used to derive physical and mental component summary scores, ranging from 0 to 100, with higher scores indicating better QOL (0=Poorest Health; 100=Best Health). Mean change from baseline = post-baseline value - baseline value; a higher value signifies improvement.
Time Frame: Baseline and Months 12, 24 and 36
Population: Randomized and transplanted participants
Measure: Mean (Standard Error); unit: units on SF-36 scale
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
units on SF-36 scale
  Physical functioning (Month 12): number analyzed (Participants) | 137 | 147 | 149
  Physical functioning (Month 12) | 2.1 (0.849) | 3.6 (0.820) | 1.9 (0.814)
  Role-physical (Month 12): number analyzed (Participants) | 138 | 147 | 149
  Role-physical (Month 12) | 5.2 (0.912) | 6.2 (0.883) | 4.7 (0.877)
  Bodily pain (Month 12): number analyzed (Participants) | 136 | 148 | 147
  Bodily pain (Month 12) | 2.9 (0.925) | 0.9 (0.887) | -0.7 (0.890)
  General health (Month 12): number analyzed (Participants) | 139 | 149 | 150
  General health (Month 12) | 2.9 (0.747) | 2.4 (0.722) | 2.1 (0.719)
  Vitality (Month 12): number analyzed (Participants) | 136 | 147 | 184
  Vitality (Month 12) | 4.1 (0.845) | 3.6 (0.814) | 2.9 (0.808)
  Social functioning (Month 12): number analyzed (Participants) | 138 | 149 | 149
  Social functioning (Month 12) | 4.2 (0.863) | 3.5 (0.830) | 2.1 (0.827)
  Role-emotional (Month 12): number analyzed (Participants) | 138 | 145 | 144
  Role-emotional (Month 12) | 2.0 (1.049) | 2.4 (1.019) | 3.5 (1.026)
  Mental health (Month 12): number analyzed (Participants) | 136 | 147 | 149
  Mental health (Month 12) | 2.7 (0.909) | 1.7 (0.875) | 2.4 (0.869)
  Physical functioning (Month 24): number analyzed (Participants) | 145 | 151 | 153
  Physical functioning (Month 24) | 1.5 (0.826) | 3.5 (0.810) | 0.7 (0.804)
  Role-physical (Month 24): number analyzed (Participants) | 145 | 150 | 151
  Role-physical (Month 24) | 5.3 (0.845) | 6.1 (0.830) | 4.3 (0.827)
  Bodily pain (Month 24): number analyzed (Participants) | 144 | 152 | 152
  Bodily pain (Month 24) | 2.0 (0.915) | 0.0 (0.891) | -1.9 (0.891)
  General health (Month 24): number analyzed (Participants) | 147 | 152 | 154
  General health (Month 24) | 2.6 (0.749) | 2.0 (0.737) | 0.6 (0.732)
  Vitality (Month 24): number analyzed (Participants) | 145 | 150 | 153
  Vitality (Month 24) | 3.9 (0.813) | 3.1 (0.801) | 1.4 (0.793)
  Social functioning (Month 24): number analyzed (Participants) | 146 | 152 | 153
  Social functioning (Month 24) | 3.2 (0.824) | 5.0 (0.807) | 2.1 (0.805)
  Role-emotional (Month 24): number analyzed (Participants) | 144 | 148 | 147
  Role-emotional (Month 24) | 2.5 (0.990) | 3.0 (0.972) | 2.9 (0.979)
  Mental health (Month 24): number analyzed (Participants) | 145 | 150 | 153
  Mental health (Month 24) | 3.0 (0.883) | 1.9 (0.869) | 1.4 (0.861)
  Physical functioning (Month 36): number analyzed (Participants) | 144 | 151 | 153
  Physical functioning (Month 36) | 1.3 (0.893) | 3.0 (0.872) | 0.7 (0.866)
  Role-physical (Month 36): number analyzed (Participants) | 144 | 148 | 152
  Role-physical (Month 36) | 5.7 (0.868) | 5.8 (0.856) | 4.1 (0.844)
  Bodily pain (Month 36): number analyzed (Participants) | 143 | 151 | 153
  Bodily pain (Month 36) | 1.6 (0.899) | 0.3 (0.875) | -2.2 (0.869)
  General health (Month 36): number analyzed (Participants) | 147 | 152 | 154
  General health (Month 36) | 2.1 (0.785) | 0.9 (0.773) | -0.5 (0.768)
  Vitality (Month 36): number analyzed (Participants) | 144 | 149 | 153
  Vitality (Month 36) | 4.1 (0.837) | 2.5 (0.823) | 1.4 (0.813)
  Social functioning (Month 36): number analyzed (Participants) | 146 | 152 | 154
  Social functioning (Month 36) | 2.9 (0.847) | 4.6 (0.830) | 1.4 (0.825)
  Role-emotional (Month 36): number analyzed (Participants) | 144 | 146 | 148
  Role-emotional (Month 36) | 2.2 (1.003) | 2.4 (0.992) | 2.5 (0.988)
  Mental health (Month 36): number analyzed (Participants) | 144 | 149 | 153
  Mental health (Month 36) | 3.6 (0.855) | 0.7 (0.841) | 0.9 (0.830)

19. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs up to 36 Months
Description: Participants with abnormal blood pressure, body weight and body temperature outside the defined normal range were graded as clinically significant vital signs by the investigator.
Time Frame: Day 1 to Month 36
Population: All randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
participants
  Heart Rate | 0 | 0 | 0
  Body Temperature | 0 | 0 | 0
  Body Weight | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities up to 36 Months
Description: Participants with laboratory values outside the defined normal range were graded as clinically significant laboratory abnormalities by the investigator. Subjects were analyzed for Alkaline phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransferase(AST), Hemoglobin, Platelet Count, Leukocytes, Bilirubin, Creatinine, Calcium, Bicarbonate, Potassium, Magnesium, Sodium, Phosphorus, Albumin, Uric Acid and Protein. Laboratory abnormalities were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3. Here 'n' signifies those subjects evaluable for this measure at specified time points for each arm, respectively.
Time Frame: Day 1 to Month 36
Population: All randomized and transplanted participants.
Measure: Number; unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
participants
  Hemoglobin (Low) (n=177,172,181) | 25 | 24 | 16
  Platelet Count (Low) (n=177,172,181) | 2 | 1 | 2
  Leukocytes (Low) (n=177,172,181) | 10 | 5 | 8
  ALP (High) (n=177,172,182) | 1 | 1 | 0
  ALT (High) (n=177,172,181) | 4 | 2 | 4
  AST (High) (n=177,172,181) | 1 | 1 | 0
  Bilirubin, Total (High) (n=177,172,182) | 0 | 2 | 1
  Creatinine (High) (n=177,172,182) | 125 | 117 | 128
  Calcium, Total (Low) (n=177,172,182) | 19 | 14 | 10
  Calcium, Total (High) (n=177,172,182) | 2 | 2 | 1
  Bicarbonate (Low) (n=176,171,181) | 2 | 1 | 2
  Bicarbonate (High) (n=176,171,181) | 0 | 0 | 0
  Potassium, Serum (Low)(n=177,172,181) | 6 | 3 | 9
  Potassium, Serum (High)(n=177,172,181) | 8 | 6 | 11
  Magnesium, Serum (Low)(n=177,172,181) | 6 | 3 | 1
  Magnesium, Serum (High)(n=177,172,181) | 6 | 4 | 9
  Sodium, Serum (Low)(n=177,172,181) | 18 | 16 | 23
  Sodium, Serum (High)(n=177,172,181) | 0 | 0 | 1
  Phosphorus (Low) (n=177,172,182) | 66 | 58 | 44
  Albumin (Low) (n=177,172,182) | 2 | 4 | 1
  Uric Acid (High) (n=177,172,182) | 31 | 34 | 60
  Protein, Urine (High) (n=173,168,177) | 44 | 37 | 43

21. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Related AEs and SAEs, AEs Leading to Discontinuation and Who Died up to Month 36
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: Day 1 to Month 36
Population: All randomized and transplanted participants
Measure: Number; unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
participants
  AEs | 182 | 174 | 184
  SAEs | 149 | 139 | 146
  AEs leading to Discontinuation | 34 | 36 | 44
  SAEs leading to Discontinuation | 31 | 31 | 28
  Related AEs | 115 | 106 | 141
  Related SAEs | 60 | 51 | 58
  Deaths | 22 | 15 | 17

22. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Related AEs and SAEs, AEs Leading to Discontinuation and Who Died up to Month 84
Description: as for outcome 21
Time Frame: Day 1 to Month 84
Population: All randomized and transplanted participants who completed 36 months of treatment and continued into long-term extension phase
Measure: Number; unit: participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 104 | 113 | 87
participants
  AEs | 104 | 113 | 87
  SAEs | 94 | 104 | 73
  AEs leading to Discontinuation | 14 | 14 | 7
  SAEs leading to Discontinuation | 94 | 104 | 7
  Deaths | 14 | 21 | 9

23. Secondary Outcome: Percentage of Participants With Graft Loss or Death to Month 84
Description: Participant and graft survival at 84 months was summarized within each treatment group.
Time Frame: Randomization to date of death, up to 84 months
Population: All randomized and transplanted participants
Measure: Number; unit: percentage of participants
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin A (CsA)
Number analyzed (Participants) | 184 | 175 | 184
percentage of participants
  Graft Loss or Death | 29.3 | 30.9 | 28.3
  Graft Loss | 11.4 | 13.1 | 15.8
  Death | 20.1 | 21.1 | 15.8
  Death with Functioning Graft | 17.9 | 17.7 | 12.5

ADVERSE EVENTS:
Time Frame: Randomization to Month 84
Groups:
- Cyclosporin (CsA): Cyclosporin A 410 mg/kg capsules, orally, twice daily in 2 divided dose for 1 month, to maintain serum concentration of 150-300 ng/mL. The subsequent dose was adjusted to maintain a predefined range of trough serum concentrations of 100-250/mL, daily for up to 84 months.
Arm/Group | Belatacept More Intensive (MI) Regimen | Belatacept Less Intensive (LI) Regimen | Cyclosporin (CsA)
Serious Adverse Events (participants affected / at risk) | 162/184 | 157/175 | 152/184
Other Adverse Events (participants affected / at risk) | 177/184 | 171/175 | 179/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept More Intensive (MI) Regimen (N=184) | Belatacept Less Intensive (LI) Regimen (N=175) | Cyclosporin (CsA) (N=184)
Abdominal hernia (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 2 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 6 | 12
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 10 | 5 | 4
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 3 | 1 | 5
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 1
Cytomegalovirus gastritis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 18 | 16 | 13
Death (General disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 4
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 8 | 3 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 2
Ileus (Gastrointestinal disorders) | 1 | 2 | 1
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Peritoneal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia cryptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 1
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 6 | 4
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Ureteric dilatation (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 4 | 3 | 4
Urinary fistula (Renal and urinary disorders) | 1 | 0 | 6
Urinary tract infection enterococcal (Infections and infestations) | 1 | 2 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 1 | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Antibody test positive (Investigations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
BK virus infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 3 | 3
Cardiogenic shock (Cardiac disorders) | 2 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral aspergillosis (Infections and infestations) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1
Chorioretinitis (Infections and infestations) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 10 | 6
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 2 | 1 | 5
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic cyst infection (Infections and infestations) | 1 | 1 | 3
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 2
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 4 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Leishmaniasis (Infections and infestations) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 3 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Oedema (General disorders) | 2 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 2
Perirenal haematoma (Injury, poisoning and procedural complications) | 2 | 3 | 1
Phlebitis (Vascular disorders) | 2 | 0 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 2
Pseudomonal sepsis (Infections and infestations) | 2 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Renal cyst infection (Infections and infestations) | 0 | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 3
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transplant dysfunction (Injury, poisoning and procedural complications) | 9 | 6 | 11
Tuberculosis of eye (Infections and infestations) | 0 | 1 | 0
Urethral disorder (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Vascular stenosis (Vascular disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 11 | 9 | 6
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1 | 1
Blood creatine increased (Investigations) | 1 | 1 | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 4
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Device malfunction (General disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 14 | 10
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 3
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 4 | 7 | 6
Haematoma (Vascular disorders) | 2 | 3 | 4
Haemorrhagic infarction (Vascular disorders) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 1 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 1 | 1
Pancreatic enzymes increased (Investigations) | 0 | 1 | 0
Perinephric effusion (Renal and urinary disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 2 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Renal infarct (Renal and urinary disorders) | 1 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 6 | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 3 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Septic shock (Infections and infestations) | 2 | 2 | 6
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 2
Strongyloidiasis (Infections and infestations) | 0 | 2 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 3 | 2
Venous thrombosis (Vascular disorders) | 0 | 3 | 0
Weight decreased (Investigations) | 0 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Angiopathy (Vascular disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cerebral fungal infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 4 | 2
Dementia (Nervous system disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dysentery (Infections and infestations) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Emphysematous cystitis (Infections and infestations) | 1 | 0 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Haemorrhagic cyst (General disorders) | 0 | 0 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Mycoplasma infection (Infections and infestations) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 7 | 3 | 3
Obstructive uropathy (Renal and urinary disorders) | 2 | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Pulmonary tuberculosis (Infections and infestations) | 3 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 3
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular atrophy (Renal and urinary disorders) | 0 | 0 | 1
Respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Sepsis (Infections and infestations) | 8 | 10 | 15
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 2
Sinusitis bacterial (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Sudden death (General disorders) | 3 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Ulcer haemorrhage (General disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Venous stenosis (Vascular disorders) | 0 | 0 | 1
Wound infection (Infections and infestations) | 2 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Abscess rupture (Infections and infestations) | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bacterial pyelonephritis (Infections and infestations) | 2 | 0 | 1
Bladder neck sclerosis (Renal and urinary disorders) | 0 | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cardiac death (General disorders) | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 6 | 1 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 2 | 1
Convulsion (Nervous system disorders) | 1 | 2 | 3
Cystitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus enteritis (Infections and infestations) | 1 | 0 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Drug intolerance (General disorders) | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 3 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 4 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 2
Human polyomavirus infection (Infections and infestations) | 0 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 3
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 4 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Polyomavirus test positive (Investigations) | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 2 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 2 | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 4 | 1 | 7
Renal artery dissection (Renal and urinary disorders) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal tubular disorder (Renal and urinary disorders) | 1 | 0 | 2
Retinal vein thrombosis (Eye disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 3
Tracheobronchitis (Infections and infestations) | 0 | 2 | 0
Uterine malposition (Reproductive system and breast disorders) | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 6
White blood cells urine positive (Investigations) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 3 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Adrenal mass (Endocrine disorders) | 0 | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 2 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 14 | 11 | 17
Blood glucose abnormal (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 3 | 4
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Chest pain (General disorders) | 5 | 3 | 4
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 4
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 2 | 1
Cytomegalovirus gastroenteritis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus syndrome (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1
Gastroenteritis (Infections and infestations) | 8 | 6 | 8
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 4 | 4 | 2
Infection (Infections and infestations) | 0 | 0 | 1
Joint tuberculosis (Infections and infestations) | 1 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Kidney infection (Infections and infestations) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 2 | 2 | 0
Mononeuropathy (Nervous system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 3
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 15 | 14 | 11
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Polyomavirus-associated nephropathy (Infections and infestations) | 3 | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 7 | 12 | 11
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Transplant abscess (Infections and infestations) | 0 | 2 | 1
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Ureteral necrosis (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 2 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 3 | 3
Urosepsis (Infections and infestations) | 6 | 7 | 6
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 4 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 | 8 | 6
Cystitis bacterial (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Disseminated cytomegaloviral infection (Infections and infestations) | 0 | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 2
Encephalitis toxic (Nervous system disorders) | 0 | 0 | 1
Encephalomyelitis (Infections and infestations) | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 1 | 0
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Escherichia test positive (Investigations) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 2 | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypertension (Vascular disorders) | 2 | 5 | 3
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0
Infected lymphocele (Infections and infestations) | 0 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 2 | 5
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Lymphocele (Vascular disorders) | 2 | 5 | 11
Macular fibrosis (Eye disorders) | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Postrenal failure (Renal and urinary disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 3 | 1
Pyelonephritis (Infections and infestations) | 12 | 6 | 14
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 4
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 1 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 3 | 9
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Renal transplant failure (Injury, poisoning and procedural complications) | 1 | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 2 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tuberculous laryngitis (Infections and infestations) | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 25 | 28 | 26
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 2
Abscess (Infections and infestations) | 3 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 4 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 3 | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 9 | 11 | 3
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Bacteraemia (Infections and infestations) | 3 | 1 | 5
Bacterial prostatitis (Infections and infestations) | 0 | 1 | 0
Brain mass (Nervous system disorders) | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 5 | 4 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Cryptococcosis (Infections and infestations) | 1 | 3 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Device related infection (Infections and infestations) | 2 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0
Extravasation (General disorders) | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0 | 0
Gangrene (Infections and infestations) | 4 | 2 | 0
Graft complication (Injury, poisoning and procedural complications) | 3 | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 3 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 3
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0
Post transplant distal limb syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 3 | 2 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Priapism (Reproductive system and breast disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Pyrexia (General disorders) | 17 | 10 | 12
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 2 | 5 | 7
Renal haemorrhage (Renal and urinary disorders) | 2 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 4 | 3 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Shock (Vascular disorders) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2
Ureteric fistula (Renal and urinary disorders) | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept More Intensive (MI) Regimen (N=184) | Belatacept Less Intensive (LI) Regimen (N=175) | Cyclosporin (CsA) (N=184)
Chills (General disorders) | 9 | 6 | 9
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 14 | 9 | 22
Conjunctivitis (Infections and infestations) | 15 | 9 | 7
Constipation (Gastrointestinal disorders) | 61 | 63 | 79
Contusion (Injury, poisoning and procedural complications) | 8 | 11 | 4
Cytomegalovirus infection (Infections and infestations) | 22 | 18 | 17
Dyslipidaemia (Metabolism and nutrition disorders) | 34 | 29 | 41
Gastritis (Gastrointestinal disorders) | 8 | 7 | 9
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1 | 9
Herpes zoster (Infections and infestations) | 21 | 17 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 21 | 20 | 23
Hyperparathyroidism (Endocrine disorders) | 7 | 5 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 12 | 13
Leukocytosis (Blood and lymphatic system disorders) | 15 | 12 | 9
Ligament sprain (Injury, poisoning and procedural complications) | 8 | 1 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 15 | 10
Abdominal distension (Gastrointestinal disorders) | 13 | 13 | 19
Bronchitis (Infections and infestations) | 37 | 36 | 25
Dehydration (Metabolism and nutrition disorders) | 13 | 10 | 8
Dyspepsia (Gastrointestinal disorders) | 22 | 16 | 20
Ecchymosis (Skin and subcutaneous tissue disorders) | 13 | 4 | 9
Escherichia urinary tract infection (Infections and infestations) | 9 | 6 | 13
Haemorrhoids (Gastrointestinal disorders) | 16 | 13 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 16 | 16 | 31
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 9
Oedema (General disorders) | 26 | 23 | 30
Proteinuria (Renal and urinary disorders) | 40 | 36 | 29
Sinusitis (Infections and infestations) | 19 | 23 | 20
Transplant dysfunction (Injury, poisoning and procedural complications) | 65 | 64 | 85
Vertigo (Ear and labyrinth disorders) | 5 | 14 | 8
Weight increased (Investigations) | 15 | 13 | 11
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 5 | 10
Abdominal pain (Gastrointestinal disorders) | 30 | 39 | 33
Anaemia (Blood and lymphatic system disorders) | 98 | 93 | 103
Aphthous stomatitis (Gastrointestinal disorders) | 10 | 13 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 56 | 41
Diarrhoea (Gastrointestinal disorders) | 103 | 94 | 74
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 40 | 37
Fatigue (General disorders) | 26 | 22 | 19
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 9
Haematoma (Vascular disorders) | 16 | 16 | 18
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 8 | 9 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 47 | 40 | 40
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 13 | 12
Incision site pain (Injury, poisoning and procedural complications) | 26 | 22 | 36
Influenza (Infections and infestations) | 17 | 16 | 18
Nasopharyngitis (Infections and infestations) | 45 | 44 | 38
Pain (General disorders) | 13 | 13 | 14
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 2 | 9
Respiratory tract infection (Infections and infestations) | 6 | 13 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 13 | 11
Tremor (Nervous system disorders) | 17 | 21 | 31
Upper respiratory tract infection (Infections and infestations) | 35 | 29 | 23
Weight decreased (Investigations) | 17 | 21 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 14 | 18 | 19
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 15 | 10 | 8
Dysuria (Renal and urinary disorders) | 25 | 23 | 16
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 9 | 9
Headache (Nervous system disorders) | 37 | 41 | 47
Hydronephrosis (Renal and urinary disorders) | 9 | 2 | 11
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 5 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 | 14 | 26
Metabolic acidosis (Metabolism and nutrition disorders) | 15 | 16 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 17 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 9 | 17
Oral herpes (Infections and infestations) | 13 | 14 | 9
Polycythaemia (Blood and lymphatic system disorders) | 4 | 10 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 8 | 6
Abdominal pain upper (Gastrointestinal disorders) | 21 | 25 | 27
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 4 | 7 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 43 | 34
Fungal skin infection (Infections and infestations) | 8 | 9 | 8
Gout (Metabolism and nutrition disorders) | 3 | 11 | 7
Haematuria (Renal and urinary disorders) | 41 | 39 | 36
Hyperkalaemia (Metabolism and nutrition disorders) | 43 | 47 | 44
Hypocalcaemia (Metabolism and nutrition disorders) | 35 | 37 | 22
Insomnia (Psychiatric disorders) | 37 | 31 | 39
Leukocyturia (Renal and urinary disorders) | 13 | 14 | 12
Osteoporosis (Musculoskeletal and connective tissue disorders) | 13 | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 35 | 34 | 42
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 18 | 6
Sinus bradycardia (Cardiac disorders) | 8 | 4 | 9
Tachycardia (Cardiac disorders) | 14 | 22 | 12
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 18
Vomiting (Gastrointestinal disorders) | 37 | 51 | 44
Wound complication (Injury, poisoning and procedural complications) | 3 | 5 | 9
Anxiety (Psychiatric disorders) | 27 | 20 | 30
Asthenia (General disorders) | 23 | 17 | 23
Blood creatinine increased (Investigations) | 29 | 29 | 31
Blood pressure increased (Investigations) | 8 | 5 | 10
C-reactive protein increased (Investigations) | 12 | 14 | 11
Chest pain (General disorders) | 22 | 24 | 24
Decreased appetite (Metabolism and nutrition disorders) | 15 | 16 | 17
Flatulence (Gastrointestinal disorders) | 5 | 5 | 10
Gastroenteritis (Infections and infestations) | 8 | 18 | 22
Hypercalcaemia (Metabolism and nutrition disorders) | 24 | 16 | 22
Hyperlipidaemia (Metabolism and nutrition disorders) | 13 | 13 | 13
Hyperphosphataemia (Metabolism and nutrition disorders) | 16 | 15 | 15
Hypotension (Vascular disorders) | 38 | 52 | 29
Left ventricular hypertrophy (Cardiac disorders) | 5 | 9 | 6
Neutropenia (Blood and lymphatic system disorders) | 12 | 10 | 12
Onychomycosis (Infections and infestations) | 14 | 6 | 8
Oral candidiasis (Infections and infestations) | 14 | 10 | 13
Peripheral swelling (General disorders) | 10 | 14 | 12
Pneumonia (Infections and infestations) | 7 | 15 | 11
Renal failure acute (Renal and urinary disorders) | 4 | 7 | 9
Urinary retention (Renal and urinary disorders) | 5 | 6 | 11
Bradycardia (Cardiac disorders) | 10 | 7 | 12
Cataract (Eye disorders) | 20 | 13 | 16
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 10 | 20 | 17
Cushingoid (Endocrine disorders) | 6 | 7 | 9
Fall (Injury, poisoning and procedural complications) | 16 | 8 | 11
Fluid overload (Metabolism and nutrition disorders) | 11 | 5 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 35 | 29 | 37
Hypertension (Vascular disorders) | 63 | 63 | 80
Hypophosphataemia (Metabolism and nutrition disorders) | 35 | 34 | 22
Leukopenia (Blood and lymphatic system disorders) | 51 | 40 | 48
Lymphocele (Vascular disorders) | 9 | 7 | 15
Oedema peripheral (General disorders) | 92 | 81 | 96
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 9 | 11
Osteopenia (Musculoskeletal and connective tissue disorders) | 10 | 7 | 6
Renal impairment (Renal and urinary disorders) | 13 | 13 | 19
Rhinitis (Infections and infestations) | 11 | 8 | 11
Sciatica (Nervous system disorders) | 7 | 11 | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 18 | 15 | 11
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 6 | 11
Urinary tract infection (Infections and infestations) | 79 | 76 | 86
Acidosis (Metabolism and nutrition disorders) | 16 | 14 | 15
Acne (Skin and subcutaneous tissue disorders) | 7 | 12 | 15
Angina pectoris (Cardiac disorders) | 5 | 8 | 12
Atrial fibrillation (Cardiac disorders) | 16 | 11 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 44 | 39
Depression (Psychiatric disorders) | 8 | 16 | 18
Dizziness (Nervous system disorders) | 26 | 18 | 18
Erectile dysfunction (Reproductive system and breast disorders) | 12 | 9 | 5
Lymphopenia (Blood and lymphatic system disorders) | 10 | 12 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 4 | 10
Nausea (Gastrointestinal disorders) | 54 | 49 | 52
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 9
Paraesthesia (Nervous system disorders) | 11 | 13 | 16
Procedural pain (Injury, poisoning and procedural complications) | 36 | 38 | 37
Pyrexia (General disorders) | 56 | 64 | 52
Renal tubular necrosis (Renal and urinary disorders) | 17 | 21 | 30
Tinea versicolour (Infections and infestations) | 2 | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less